CLINICAL TRIAL: NCT00981838
Title: A Prospective, Sequential Study to Assess the Efficacy of Rituximab Therapy in Maintaining Remission of Nephrotic Syndrome After Steroid and Immunosuppressive Therapy Withdrawal in Patients With Steroid-dependant or Multirelapsing Minimal Change Disease or Focal Segmental Glomerulosclerosis (NEMO Study)
Brief Title: Rituximab in Multirelapsing Minimal Change Disease (MCD) or Focal Segmental Glomerulosclerosis (FSGS)
Acronym: NEMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEMO; 2008-006750-17 (EudraCT Number)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Rituximab (375 mg/m2).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab (375 mg/m2) will be given as a single intravenous infusion after reconstitution in normal saline to a concentration of 1 mg/ml given though a 0.22 micron in line filter. The initial infusion rate will be 1 ml/kg/h and will be progressively increased up to 4 ml/kg/h according to drug tolerability. Pre-medication with steroids and/or antihistaminic agents will be done according to per-center's practice.Rituximab administration will be repeated in those patients > 5 B cells/mm3 in the peripheral blood on the day after first Rituximab administration.

SUMMARY:
Background. Patients, especially children, with steroid-dependent or multirelapsing nephrotic syndrome (NS) secondary to minimal change disease (MCD) or idiopathic focal and segmental glomerulosclerosis (FSGS) on continuous treatment with steroids and/or other immunosuppressive agents to limit or prevent recurrences are at increased risk of severe drug-related adverse events. Case reports suggest that Rituximab, a B cell depleting monoclonal antibody, could be a safe and effective alternative to steroid or immunosuppressants to achieve and maintain remission in this population.

Objectives. The study is primarily aimed at evaluating whether Rituximab may maintain stable NS remission after tapering and withdrawal of steroid and immunosuppressive therapy in patients with MCD or FSGS and steroid-dependent or multirelapsing NS. Secondarily, the study will assess whether Rituximab allows reducing maintenance doses of steroids and other immunosuppressants (in those who relapse), thus limiting treatment related side effects and costs.

Methods. This prospective, sequential, open, study will include 20 patients with histology evidence of MCD or FSGS and steroid-dependant or multirelapsing NS, who are on stable complete or partial remission since at least 1 month and, based on their previous history, are expected to invariably relapse after steroid/immunosuppression withdrawal. After baseline evaluation of clinical, laboratory and kidney function parameters [including glomerular filtration rate (GFR), renal plasma flow (RPF), albumin and sodium fractional clearance and the glomerular albumin permeability assay (Palb)], patients will receive one Rituximab infusion that will be repeated 1 week later if CD20 cells are not fully depleted from the circulation. Then ongoing immunosuppression will be progressively tapered up to complete withdrawal over 6 to 9 months. 24h proteinuria will be monitored monthly and spot urine will be tested daily by albustix to early detect disease relapses. Baseline evaluations will be repeated at study end (1 year). Relapses will be treated with high-dose steroids as per center practice and the last immunosuppressive therapy effective in preventing disease reactivation will be reintroduced.

Expected results. Rituximab is expected to prevent NS recurrence following tapering and discontinuation of steroid and other immunosuppressants. Maintaining remission without chronic immunosuppression is expected to minimize risks and costs of therapy and to remarkably improve patient outcomes.

DETAILED DESCRIPTION:
BACKGROUND Nephrotic syndrome (NS)affects 2 every 100,000 children younger than 16 years. Minimal change disease (MCD) accounts for around 90 percent of cases and most of the remaining ones are associated with focal segmental glomerulosclerosis (FSGS). Patients with NS are at increased risk for life-threatening infections and thromboembolic episodes, and are often affected by dyslipidemia and osteoporosis. Glucocorticoids are first-line treatment and may achieve remission in about 90% of patients with MCD and in 20 to 60% of those with FSGS. In about 20% to 60% of those achieving remission, however, steroid withdrawal is followed by a recurrence of the disease. These patients require chronic steroid therapy (steroid-dependent cases): this prevents relapses in most cases but is invariably associated with severe adverse effects including growth retardation, infections, malignancies, hypertension, impaired glucose tolerance, weight gain and somatic changes. In a small proportion of patients, recurrences occur even under chronic steroid therapy (multirelapsing cases). In these cases, several approaches have been used to control disease activity including plasmapheresis and add-on therapy with cyclophosphamide, cyclosporine, mycophenolate mofetil and other immunosuppressants. Chronic immunosuppression, however, seldom achieves persistent remission and is invariably burdened by serious adverse effects including gonadotoxicity and sterility, opportunistic infections, malignancies, bone marrow depression and renal toxicity. Thus, safer and more effective treatments are urgently needed for these patients.

Rituximab, a chimeric monoclonal antibody targeted to the CD20 antigen of B cells able to induce antibody-dependent and complement-mediated lysis of these cells, has been reported to be effective in children with NS secondary to MCD or FSGS unresponsive to other immunosuppressive treatments. Rituximab achieved persistent NS remission in a patient with MCD diagnosed at age of 30 yrs who had a history of frequent relapses refractory to treatment with other immunosuppressants. Thus, chronic MCD persisting into adult-years may respond to rituximab and sustained remissions are possible despite long-term disease and after other treatments have failed. Along the same line, rituximab achieved prompt and persistent remission in an adult with steroid and mycophenolate mofetil-resistant MCD and in two patients with FSGS and steroid-resistant NS.

The above findings suggest that rituximab may have a role in the treatment of patients who require chronic exposure to steroids and/or other immunosuppressants to prevent or limit disease reactivation. Thus, main goal of the present study is to assess whether rituximab administration may allow tapering and withdrawing ongoing treatment without exposing the patients to the risk of disease recurrence.

AIMS Primary

* To evaluate whether Rituximab therapy is able to prevent NS recurrence after complete withdrawal of steroids and other immunosuppressive treatments in patients with steroid-dependant or multirelapsing NS on sustained remission for at least 1 month.

Secondary

* To assess whether Rituximab therapy may reduce the need for steroids and other immunosuppressive agents to prevent and treat further disease relapses;
* To evaluate whether tapering or withdrawal of immunosuppressant therapy is associated with regression of the related toxicities, such as growth retardation, hypertension, impaired glucose tolerance and dyslipidemia;
* To assess whether persistent NS remission is associated with an improvement of kidney function and of renal hemodynamics;
* To study whether proteinuria remission is associated with the disappearance of albumin permeability factor(s) from patient's sera;
* To assess the safety profile of the rituximab treatment;
* To evaluate the cost/effectiveness of the study treatment.

ELIGIBILITY:
Inclusion criteria:

* Males and females
* Steroid-dependent or multirelapsing NS (defined on the basis of the occurrence of more than 2 relapses in the previous year in spite of steroid and/or other immunosuppressive therapy). Only patients reported to invariably relapse upon treatment tapering or withdrawal who are on stable (from at least 1 month) complete (<0.3 g/24h for adults or <4 mg/h/m2 for children) or partial (<3.5 g/24h for adults or <40 mg/h/m2 for children) remission of the NS will be included;
* Histological diagnosis of MCD or FSGS or mesangial proliferative GN;
* Written informed consent (or consent from parents or tutors for underage patients).

Exclusion criteria:

* Advanced renal failure (creatinine clearance less than 20 ml/min/1.73m2);
* Evidence of B or C virus infection;
* Refractory or persistent NS;
* Genetic mutations associated with intrinsic abnormalities of the glomerular barrier that would hardly be affected by rituximab treatment;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity;
* Evidence of an uncooperative attitude;
* Previous diagnosis of: intellectual disability/mental retardation, dementia, schizophrenia.
* Any evidence that patient will not be able to complete the trial follow-up.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of NS. | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 month.

SECONDARY OUTCOMES:
The dose of immunosuppressive therapy to prevent further NS relapses. Adverse effects of immunosuppressive therapy, such as arterial hypertension and need for antihypertensive therapy, impaired glucose tolerance, dyslipidemia, renal dysfunction. Kidney | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Study Chair — Mario Negri Institute for Pharmacological Research
Locations (7):
- Italy (7):
  - Hospital "Azienda Ospedaliera Ospedali Riunitidi Bergamo"Unit of Nephrology and Dialysis, Bergamo, Bergamo
  - Hospital "Azienda Ospedaliera santobono-Pausilipon" - Unit of Nephrology and Dialysis, Napoli, Napoli
  - Hospital "Azienda Ospedaliero Universitaria Federico II" - Nephrology, Napoli, Napoli
  - Hospital "Seconda Università di Napoli" - Policlinico Nuovo, Napoli, Napoli
  - Hospital "IRCCS Pediatrico Bambino Gesù di Roma" - Department of Nephrology and Pediatric Urology, Roma, Roma
  - Hospital "IRCCS Istituto per l'Infanzia Burlo Garofolo" - Pediatric Nephrology Service, Trieste, Trieste
  - Hospital "Ospedale di Cattinara" - Ambulatory of nephrology, Trieste, Trieste

REFERENCES:
- [Derived] Ruggenenti P, Ruggiero B, Cravedi P, Vivarelli M, Massella L, Marasa M, Chianca A, Rubis N, Ene-Iordache B, Rudnicki M, Pollastro RM, Capasso G, Pisani A, Pennesi M, Emma F, Remuzzi G; Rituximab in Nephrotic Syndrome of Steroid-Dependent or Frequently Relapsing Minimal Change Disease Or Focal Segmental Glomerulosclerosis (NEMO) Study Group. Rituximab in steroid-dependent or frequently relapsing idiopathic nephrotic syndrome. J Am Soc Nephrol. 2014 Apr;25(4):850-63. doi: 10.1681/ASN.2013030251. Epub 2014 Jan 30. PMID 24480824